CLINICAL TRIAL: NCT06392464
Title: Clinical Validation Study of Naevia Medical, a Clinical Decision Support System, in Heart Valve Disease
Brief Title: Validation of Naevia Medical in Valvulopathies
Acronym: CDSS-Valve
Status: Completed | Type: Observational
Sponsor: Dilemma Solutions S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024/104
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Results first posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Heart Valve Disease
Keywords: clinical decision support system; artificial intelligence; cdss
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with heart valve disease: The same group of patients is evaluated with a pre-test-post-test design with a randomly assigned group, utilizing a longitudinal approach with repeated measures and retrospective validation.
  Interventions: Device: Clinical decision support system (software)

INTERVENTIONS:
Device: Clinical decision support system (software) — Use of a clinical decision support system. "Naevia Medical" is clinical decision support software (CDSS) that, based on clinical input data (patient history, symptoms, complementary test data, etc.) from adult patients with heart disease, provides healthcare professionals with prioritized, justified, and referenced recommendations and knowledge-related suggestions related to diagnosis, prognosis, and/or treatment (recommended tests, medications, alerts, etc.)

SUMMARY:
The study aims to validate naevia medical, a knowledge-based clinical decision support system (CDSS), for clinical benefit and safety in cases of cardiac valvulopathies. Using a series of retrospective clinical cases of heart valve disease, the research will evaluate the number of appropriate and inappropriate recommendations during baseline measurement (conventional management) and after CDSS activation.

DETAILED DESCRIPTION:
The objective of this study is to validate both the clinical benefit and safety of a knowledge-based clinical decision support system (CDSS), naevia medical, applied to clinical cases of cardiac valvulopathies.

naevia medical aims to bridge the gap between scientific evidence and medical practice by improving adherence to scientific recommendations.

The research aims to establish and verify that the naevia medical product is suitable for its intended purposes and provides the specified intended functionality as outlined by its manufacturer under normal conditions of use. It seeks to verify the clinical benefits of the product compared to conventional management by enhancing healthcare professionals' ability to provide a greater number of scientifically based recommendations tailored to each patient's specific situation. Additionally, the study aims to establish the clinical safety of the product by identifying potential undesirable side effects under normal usage conditions and evaluating whether these effects constitute acceptable risks in relation to the benefits provided.

To achieve these objectives, a clinical research study will be conducted to assess naevia medical's capacity to increase appropriate recommendations and decrease inappropriate recommendations received by patients with valvulopathy, compared to conventional management without support.

The study proposes a pre-test-post-test design with a randomly assigned group, utilizing a longitudinal approach with repeated measures and retrospective validation. Evaluation criteria will focus on the number of appropriate and inappropriate recommendations during baseline measurement (conventional management) and after CDSS activation, using a series of retrospective clinical cases of heart valve disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients randomly selected from those presented during the year 2022 in medical-surgical sessions, with a primary diagnosis of:

  * aortic valve stenosis
  * aortic insufficiency
  * mitral valve stenosis
  * mitral insufficiency (greater than moderate severity)..
* Patients randomly selected from valvulopathy clinic records attended during the year 2022, with a primary diagnosis of

  * aortic valve stenosis
  * aortic insufficiency
  * mitral valve stenosis
  * mitral insufficiency (greater than moderate severity)

Exclusion Criteria:

* Subjects under 18 years old.
* Inability to anonymize the case.
* Clinical cases of valvulopathies in which a complex congenital heart disease coexists.
* Clinical cases that do not meet the minimum data set necessary for decision-making.
* Clinical cases with a primary diagnosis other than valvulopathy.
* Presence of bacterial endocarditis

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients evaluated in the outpatient clinic affected by heart valve disease
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Official webpage of the product — https://naeviamedical.com/en/index/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The same group of 106 cases was evaluated before and after the CDSS activation.
Groups:
- Patients With Heart Valve Disease: The same group of patients is evaluated with a pre-test-post-test design with a randomly assigned group, utilizing a longitudinal approach with repeated measures and retrospective validation.
  The clinical management of the included cases was retrospectively evaluated by a panel of 3 experts with access to the most updated guidelines, without activating the CDSS.
Period: Overall Study
Arm/Group | Patients With Heart Valve Disease
Started (The same group of 106 cases was evaluated with and without the CDSS activation) | 106 (The same group of 106 cases was evaluated with and without the CDSS activation)
Pre-test | 106
Post-test | 106
Completed | 106 (The same group of 106 cases was evaluated with and without the CDSS activation)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 106 clinical cases of aortic stenosis, aortic insufficiency, mitral stenosis, and mitral insufficiency were selected with stratified random sampling. The conventional clinical management was retrospectively evaluated by three expert cardiologists using updated guidelines.
Arm/Group | Patients With Heart Valve Disease
Number analyzed (Participants) | 106
Age, Continuous [Mean (Full Range); unit: Years] | 73.35 [40 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 64
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Relevant Appropriate Recommendations
Description: Number of relevant appropriate recommendations. Only high-level recommendations (class I and IIa) were included and evaluated in the study.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: Recommendations
Groups:
- Patients with heart valve disease (pre-test); Patients with heart valve disease (post-test): The same group of patients is evaluated with a pre-test-post-test design with a randomly assigned group, utilizing a longitudinal approach with repeated measures and retrospective validation.
  The clinical management of the included cases was retrospectively evaluated by a panel of 3 experts with access to the most updated guidelines, without activating the CDSS.
Arm/Group | Patients with heart valve disease (pre-test) | Patients with heart valve disease (post-test)
Number analyzed (Participants) | 105 | 105
Recommendations | 2.35 (1.97) | 6.20 (2.57)

2. Primary Outcome: Number of Inappropriate Recommendations
Description: Number of inappropriate recommendations (that do not apply to the specific case)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: Recommendations
Arm/Group | Patients with heart valve disease (pre-test) | Patients With Heart Valve Disease (post-test)
Number analyzed (Participants) | 105 | 105
Recommendations | 0.29 (0.60) | 0.07 (0.29)

3. Primary Outcome: Number of Relevant Missing Recommendations
Description: Number of relevant missing recommendations. Only high-level recommendations (class I and IIa) were included and evaluated in the study.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: Recommendations
Groups:
- Patients with heart valve disease (post-test): The same group of patients is evaluated with a pre-test-post-test design with a randomly assigned group, utilizing a longitudinal approach with repeated measures and retrospective validation.
  The clinical management of the included cases was retrospectively evaluated by a panel of 3 experts with access to the most updated guidelines, with the CDSS activation.
Arm/Group | Patients with heart valve disease (pre-test) | Patients with heart valve disease (post-test)
Number analyzed (Participants) | 105 | 105
Recommendations | 3.80 (2.27) | 0.49 (0.67)

ADVERSE EVENTS:
Time Frame: N/A (retrospective evaluation)
Description: This study is a retrospective evaluation of historical cases by an expert panel assessment. The evaluation was performed with and without the activation of the CDSS. The clinical recommendations provided with conventional management and after the CDSS activation were counted and evaluated, but no new interventions were applied. Therefore, no adverse events were prospectively collected and the number of participants 'at risk' for adverse-event monitoring is 0.
Arm/Group | Patients With Heart Valve Disease
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The main limitation of the present study is its retrospective design, which does not allow to evaluate naevia's impact on clinical decision making in real life. This aspect will be addressed in further prospective studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT06392464/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT06392464/SAP_001.pdf